CLINICAL TRIAL: NCT06165809
Title: A Phase I Study to Evaluate the Safety and Tolerance of TQB3015 Tablets With Advanced Malignant Cancer.
Brief Title: A Clinical Trial of TQB3015 Tablets in Patients With Advanced Malignant Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The sponsor voluntarily withdraw the project.
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3015-I-01
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Advanced Malignant Neoplasm

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3015 tablets (Experimental): TQB3015 tables is administered as a single dose or multiple dose, 2-40mg once a day; Oral administration on fast condition, 21 days as a cycle.
  Interventions: Drug: TQB3015 tablets

INTERVENTIONS:
Drug: TQB3015 tablets — TQB3015 is a protein inhibitor

SUMMARY:
This study is divided into two stages: dose escalation and dose extension, including a single dose and a multiple dose clinical study. This is a single-center, open, non randomized, single arm study to the safety and tolerability of TQB3015 tables in patients with advanced malignant cancer.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study;
* Age: 18 to 75 years old; an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Advanced malignant tumors confirmed by tissue or cellular pathology and the routine standard treatment was ineffective or lack of effective treatment plans, or patients cannot tolerate the standard treatment;
* Has at least one assessable lesion according to Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 criteria;
* The main organs function well;
* Female patient had no plans to become pregnant and voluntarily took effective contraceptive measures during the study period and until at least 6 months after the last dose of study drug.

Exclusion Criteria:

* Concomitant disease and medical history:

  1. There were other malignant tumors occured within 3 years before the first dose of study drug.
  2. Has multiple factors affecting oral medication;
  3. Unalleviated toxicity ≥ grade 1 according to CTCAE v5.0 due to any previous therapy, excluding hair loss;
  4. Major surgical treatment, open biopsy and obvious traumatic injury were performed within 28 days before the study, or have not fully recovered from previous surgery, or are expected to require major surgical surgery during the study period;
  5. Arteriovenous thrombotic events occurred within 6 months before the first dose, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis and pulmonary embolism;
  6. Have a history of psychotropic drug abuse and can not quit or have mental disorders;
  7. Subjects with any severe and/or uncontrolled disease including active hepatitis, immunodeficiency;
* Tumor-related symptoms and treatment:

  1. Has known symptomatic central nervous system metastases and/or cancerous meningitis;
  2. Have received surgery, chemotherapy, radiation therapy (2 weeks for brain radiation therapy) or other anti-cancer therapies within 4 weeks prior to the first dose.
  3. Thoracic/abdominal/pericardial effusion with clinical symptoms or requiring repeated drainage, or drainage for the purpose of receiving treatment within one month after receiving the investigational drug for the first time.
  4. Has Participated in other clinical trials within 4 weeks before first dose.
* According to the judgement of the investigators, there are other factors that may lead to the termination of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | At the end of Cycle 1 (Day 21).
  DLT will be defined as toxicities that meet pre-defined severity criteria according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 toxicity, and assessed as having a suspected relationship to study drug that occurred from the first dose to the end of the first treatment cycle.
Maximum tolerated dose (MTD) | At the end of Cycle 1 (Day 21).
  MTD was defined as the highest dose at which dose-limiting toxicity (DLT) occurred in less than 33% of patients.
Recommended Phase II Dose (RP2D) | Baseline up to 24 months
  DLT describes side effects of a drug or other treatment that are serious enough to evaluate RP2D of TQB3015 tablets in adult patients with Advanced Malignant Cancer.
Incidence of abnormal clinical laboratory | 30 days after the last administration.
  Incidence of participants with clinical laboratory abnormalities

SECONDARY OUTCOMES:
Adverse events (AE) | 30 days after the last administration.
  The occurrence of all adverse events (AE).
Serious adverse events (SAE) | 30 days after the last administration.
  The occurrence of all serious adverse events (SAE).
Time to reach maximum (peak) plasma concentration (Tmax) | Pre-dose, at 0.5, 1, 2, 3,4, 6, 8, 11, 24, 48, 72 hours after single administration dose. Pre-dose on Cycle 1 Day 7,Cycle 1 Day 14, Cycle 1 Day21; 0.5, 1, 2, 3, 4, 6, 8, 11, 24 hours after-dose on Cycle 1 Day 21. Each cycle is 21 days.
  To characterize the pharmacokinetics of TQB3015 by assessment of time to reach maximum plasma concentration after single and multiple dosing.
Peak concentration (Cmax) | Pre-dose, at 0.5, 1, 2, 3,4, 6, 8, 11, 24, 48, 72 hours after single administration dose. Pre-dose on Cycle 1 Day 7,Cycle 1 Day 14, Cycle 1 Day21; 0.5, 1, 2, 3, 4, 6, 8, 11, 24 hours after-dose on Cycle 1 Day 21. Each cycle is 21 days.
  The maximum observed plasma concentration of study drug.
Half-life (t1/2) | Pre-dose, at 0.5, 1, 2, 3,4, 6, 8, 11, 24, 48, 72 hours after single administration dose. Pre-dose on Cycle 1 Day 7,Cycle 1 Day 14, Cycle 1 Day21; 0.5, 1, 2, 3, 4, 6, 8, 11, 24 hours after-dose on Cycle 1 Day 21. Each cycle is 21 days.
  The time required for half of the drug to be eliminated from the plasma.
Area under the concentration-time curve from zero to infinity (AUC0-∞) | Pre-dose, at 0.5, 1, 2, 3,4, 6, 8, 11, 24, 48, 72 hours after single administration dose. Pre-dose on Cycle 1 Day 7,Cycle 1 Day 14, Cycle 1 Day21; 0.5, 1, 2, 3, 4, 6, 8, 11, 24 hours after-dose on Cycle 1 Day 21. Each cycle is 21 days.
  To characterize the pharmacokinetics of TQB3015 by assessment of area under the plasma concentration time curve from 0 extrapolated to infinity.
Area under the concentration-time curve from zero to last observation (AUC [0-t]) | Pre-dose, at 0.5, 1, 2, 3,4, 6, 8, 11, 24, 48, 72 hours after single administration dose. Pre-dose on Cycle 1 Day 7,Cycle 1 Day 14, Cycle 1 Day21; 0.5, 1, 2, 3, 4, 6, 8, 11, 24 hours after-dose on Cycle 1 Day 21. Each cycle is 21 days.
  To characterize the pharmacokinetics of TQB3015 by assessment of area under the plasma concentration time curve from the first dose to a certain time point.
Apparent clearance (CL/F) | Pre-dose, at 0.5, 1, 2, 3,4, 6, 8, 11, 24, 48, 72 hours after single administration dose. Pre-dose on Cycle 1 Day 7,Cycle 1 Day 14, Cycle 1 Day21; 0.5, 1, 2, 3, 4, 6, 8, 11, 24 hours after-dose on Cycle 1 Day 21. Each cycle is 21 days.
  Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the body.
Apparent volume of distribution (Vd/F) | Pre-dose, at 0.5, 1, 2, 3,4, 6, 8, 11, 24, 48, 72 hours after single administration dose. Pre-dose on Cycle 1 Day 7,Cycle 1 Day 14, Cycle 1 Day21; 0.5, 1, 2, 3, 4, 6, 8, 11, 24 hours after-dose on Cycle 1 Day 21. Each cycle is 21 days.
  Apparent volume of distribution of the TQB3015 in plasma.
Objective response rate (ORR) | From date of the first dose until the date of first documented progression or date of death from any cause, assessed up to 100 weeks.
  The percentage of patients with complete response (CR) and/or partial response (PR) assessed by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Harbin Medical University Cancer Hospital, Harbin, Heilongjiang, China